CLINICAL TRIAL: NCT05319483
Title: The Clinical, Epidemiological and Treatment Characteristics of Head and Neck Cancer Patients Presenting to Different Levels of the Health Care System
Brief Title: The Clinical, Epidemiological and Treatment Characteristics of Head and Neck Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: 8850 PTE 2021
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Waiting Times, Patient Pathways, Effect of Lifestyle-related, Clinical and Demographic Parameters on Outcomes
Keywords: Head and neck cancer, Survival, Waiting times, Patient pathways
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention.

SUMMARY:
The aim of our study is to prospectively collect information regarding (1) the demographic, lifestyle-related and clinical characteristics of patients with head and neck cancer and (2) the waiting times to diagnosis and therapy, and the 1-, 3- and 5-year survival of patients. We plan to gain insight into the characteristics and pathways of head and neck cancer patients in Baranya County, which can in turn help to identify factors that lead to improved or worse disease outcomes. (Thus, these factors can subsequently eliminated or lessened to improve the outcome of head and neck cancer patients. )

DETAILED DESCRIPTION:
The aim of our study is to prospectively collect information regarding (1) the demographic, lifestyle-related and clinical characteristics of patients (including initial symptoms) with head and neck cancer and (2) the patient pathways and waiting times to diagnosis and therapy, the 1-, 3- and 5-year survival, and time to metastasis of patients.

Study design:

Prospective data collection and analysis, based on data collected from the clinic's electronic eMedSol database and questionnaire (regarding demographic, lifestyle and patient pathway-related data) filled in by interviewing patient.

We plan to monitor lifestyle parameters of patients (such as oral hygiene, alcohol consumption and smoking, the knowledge of patients about risk factors of head and neck cancers,etc) and clinical parameters such as time and type of first symptom, ECOG state, comorbidities, clinical stage, diagnostic workups, etc. at predetermined time intervals (upon first ENT presentation, and at 3-, 6-, 12-, and 24 month intervals.

Disease progression (time to metastasis) and overall survival will be assessed at the given time points.

By gathering data and gaining insight into the characteristics, pathways and survival of head and neck cancer patients we aim to identify factors that may lead to improved or worse disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or over presenting with head and neck cancer (with morphology of squamocellular carcinoma), who are subsequently given one of the following ICD-10 codes: Malignant neoplasms of lip, oral cavity and pharynx (C00-C14), Malignant neoplasm of larynx (C32) and for whom this is their first cancer.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria and patients who meet the inclusion criteria but for whom this is a second or recurrent cancer (they already have an "ICD-C" code) are excluded from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients 18 years or over with primary head-neck cancer (with morphology of squamocellular carcinoma, ICD codes: C00-C14, C32) and no previously documented cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of patient pathways | 2021-2024
  Initial symptoms, waiting times to diagnosis and treatment, type of healthcare provision
Lifestyle-related factors | 2021-2026
  The effects of demographic and lifestyle-related factors on clinical outcome(s) using follow-up data
Hard endpoint outcomes: Overall survival, time to metastasis, disease-free survival | 2021-2029
  Assessment of overall survival, time to metastasis, disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pécs, Clinical Centre, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No